CLINICAL TRIAL: NCT01773603
Title: Blastocyst Culture Using Time-lapse in Good Prognosis IVF Patients and Elective Single Embryo Transfer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No statistical difference observed for outcomes.
Sponsor: Dr. Murat Çetinkaya (Other)
Responsible Party: Sponsor-Investigator, Dr. Murat Çetinkaya, R&D Laboratory Manager, Memorial Sisli Hospital, Istanbul
Organization: Memorial Sisli Hospital, Istanbul (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: MC0405; IMH2013-1 (Other: Sisli Memorial Hospital)
Record Dates: First submitted 2013-01-18; First posted 2013-01-23 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Infertility
Keywords: Time-lapse; morphokinetics; blastocyst transfer; eSET
MeSH Terms: conditions — Infertility | interventions — Fetoscopes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional incubation (No Intervention): Five-day embryo culture in conventional incubators
- Embryoscope (Active Comparator): Five-day embryo culture in embryoscope which is an incubator with a built-in camera
  Interventions: Device: Embryoscope

INTERVENTIONS:
Device: Embryoscope — Five-day embryo culture in embryoscope which is an incubator with a built-in camera
  Other Names: Time-lapse monitoring of human embryos in Embryoscope
  Arms: Embryoscope

SUMMARY:
Choosing the best embryo for transfer has become the major challenge in in vitro fertilization (IVF). Morphology alone is obviously not enough and time-lapse incubation has added embryo development kinetics as another selection criterion.

This study was designed to select for the top blastocyst to be replaced, while increasing the pregnancy chance, with the local legislation regulating the number of embryos to be transferred and to establish a morphokinetic standard to be used in our clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* patients in their first or second ART treatment cycle
* no recurrent spontaneous abortions
* age<35 years
* BMI<28 kg/m2
* ≥8 oocytes retrieved

Exclusion Criteria:

* severe endometriosis
* polycystic ovary syndrome
* hydrosalpynx
* uterine pathology
* severe male factor (presenting less than 5 million motile sperm cells in total in the ejaculate)
* very severe morphological sperm defects (mainly globozoospermic or macrocephalic samples)

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2011-12; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Blastocyst formation rate | 5th day of embryonic development

SECONDARY OUTCOMES:
Clinical pregnancy rate | 7th week of pregnancy
  Clinical pregnancy was defined as the presence of a gestational sac detected on ultrasound 3 weeks after the first βhCG test, which was performed 14 days after oocyte retrieval.

CONTACTS AND LOCATIONS:
Overall Officials: Semra Kahraman, MD, Prof, Study Director — Sisli Memorial Hospital
Locations (1):
- Sisli Memorial Hospital, Istanbul, Turkey (Türkiye)